CLINICAL TRIAL: NCT05103787
Title: Impact of Bilateral Deep Parasternal Intercostal Plane Block on Intraoperative Opioid Consumption in Open Heart Surgery: a Prospective, Double-blind Randomized Controlled Study
Brief Title: Impact of Bilateral Deep Parasternal Intercostal Plane Block on Intraoperative Opioid Consumption in Open Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Aida Rosita Tantri, Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUAnes119
Record Dates: First submitted 2021-09-27; First posted 2021-11-02 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: Opioid Use
Keywords: regional anesthesia; intercostal plane block; opioid; open heart surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- deep parasternal plane block (Active Comparator): Subjects will receive bilateral deep parasternal intercostal plane block after induction of anesthesia.
  Interventions: Procedure: deep parasternal intercostal plane block; Procedure: control
- control (Placebo Comparator): subjects will receive skin puncture with needle on the same location as the treatment group without administration of local anesthetics after induction of anesthesia,
  Interventions: Procedure: deep parasternal intercostal plane block; Procedure: control

INTERVENTIONS:
Procedure: deep parasternal intercostal plane block — Twenty milliliters of 0.25% bupivacaine will be placed bilaterally in the fascial plane between internal intercostal muscle and transversus thoracis muscle at intercostal space 4 or 5, lateral from sternum, with ultrasound guidance using high-frequency linear transducer.
Procedure: control — Skin puncture with needle will be performed on the same location as the treatment group without administration of local anesthetics.

SUMMARY:
This study aims to assess the impact of bilateral deep parasternal intercostal plane block on intraoperative opioid consumption in open heart surgery

DETAILED DESCRIPTION:
High-dose opioid is associated with various side effects such as nausea, vomiting, urinary retention, and respiratory depression. The neuraxial block (intrathecal, epidural) and peripheral nerve block are regional anesthesia techniques which have the potential to reduce intraoperative opioid consumption. The deep parasternal intercostal plane block is fascial plane block which intended to block anterior cutaneous branch of intercostal nerves.

This study is a double-blind randomized controlled trial. Thirty subjects will be recruited with consecutive sampling method. Eligible subjects with signed informed consent will be randomized into two groups. The first group is the treatment group who will receive bilateral deep parasternal intercostal plane block after induction of anesthesia and the second group will be the control group who will not receive any regional anesthesia. After surgery, extubation time, adverse event (nausea, vomiting), and intensive care unit length of stay will be recorded for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* Elective open-heart surgery with median sternotomy approach

Exclusion Criteria:

* Patient who refuses to participate
* Patient with local infection in the block area
* Patient with chronic pain
* Patient with history of chronic analgesics use
* Patient who is contraindicated for local anesthetics
* Patient with cognitive disorder
* Patient with severe psychiatric disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-04-04 (Estimated); Study Completion 2022-07-04 (Estimated)

PRIMARY OUTCOMES:
Total intraoperative fentanyl dose | intraoperatively
  Total intraoperative fentanyl dose will be calculated after surgery

SECONDARY OUTCOMES:
Time to first intraoperative fentanyl | intraoperatively
  Investigators will record time to first fentanyl dose after incision
extubation time | Up to 72 hours after surgery
  Investigators will record time to extubation after surgery
opioid side effects | within 24 hours after surgery
  Incidence of nausea and vomiting
Intensive care unit length of stay | Up to 7 days after surgery
  Investigators will record total time from intensive care unit admission until patient transferred to surgical wars

CONTACTS AND LOCATIONS:
Overall Officials: Aida Rosita R Tantri, Principal Investigator — Indonesia University
Locations (2):
- Indonesia (2):
  - Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta
  - Universitas Indonesia, Central Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aydin ME, Ahiskalioglu A, Ates I, Tor IH, Borulu F, Erguney OD, Celik M, Dogan N. Efficacy of Ultrasound-Guided Transversus Thoracic Muscle Plane Block on Postoperative Opioid Consumption After Cardiac Surgery: A Prospective, Randomized, Double-Blind Study. J Cardiothorac Vasc Anesth. 2020 Nov;34(11):2996-3003. doi: 10.1053/j.jvca.2020.06.044. Epub 2020 Jun 18. PMID 32665179
- [Result] Cardinale JP, Latimer R, Curtis C, Bukovskaya Y, Kosarek L, Falterman J, Tatum DM, Trusheim J. Incorporation of the Transverse Thoracic Plane Block Into a Multimodal Early Extubation Protocol for Cardiac Surgical Patients. Semin Cardiothorac Vasc Anesth. 2021 Dec;25(4):301-309. doi: 10.1177/1089253220957484. Epub 2020 Sep 9. PMID 32907499
- [Result] Chin KJ. An Anatomical Basis for Naming Plane Blocks of the Anteromedial Chest Wall. Reg Anesth Pain Med. 2017 May/Jun;42(3):414-415. doi: 10.1097/AAP.0000000000000575. No abstract available. PMID 28419049
- [Result] Bloc S, Perot BP, Gibert H, Law Koune JD, Burg Y, Leclerc D, Vuitton AS, De La Jonquiere C, Luka M, Waldmann T, Vistarini N, Aubert S, Menager MM, Merzoug M, Naudin C, Squara P. Efficacy of parasternal block to decrease intraoperative opioid use in coronary artery bypass surgery via sternotomy: a randomized controlled trial. Reg Anesth Pain Med. 2021 Aug;46(8):671-678. doi: 10.1136/rapm-2020-102207. Epub 2021 May 14. PMID 33990437
- [Result] Vilvanathan S, Saravanababu MS, Sreedhar R, Gadhinglajkar SV, Dash PK, Sukesan S. Ultrasound-guided Modified Parasternal Intercostal Nerve Block: Role of Preemptive Analgesic Adjunct for Mitigating Poststernotomy Pain. Anesth Essays Res. 2020 Apr-Jun;14(2):300-304. doi: 10.4103/aer.AER_32_20. Epub 2020 Oct 12. PMID 33487833
- [Result] Probst S, Cech C, Haentschel D, Scholz M, Ender J. A specialized post anaesthetic care unit improves fast-track management in cardiac surgery: a prospective randomized trial. Crit Care. 2014 Aug 15;18(4):468. doi: 10.1186/s13054-014-0468-2. PMID 25123092
- [Result] Wong WT, Lai VK, Chee YE, Lee A. Fast-track cardiac care for adult cardiac surgical patients. Cochrane Database Syst Rev. 2016 Sep 12;9(9):CD003587. doi: 10.1002/14651858.CD003587.pub3. PMID 27616189
- [Result] Chakravarthy M. Regional analgesia in cardiothoracic surgery: A changing paradigm toward opioid-free anesthesia? Ann Card Anaesth. 2018 Jul-Sep;21(3):225-227. doi: 10.4103/aca.ACA_56_18. No abstract available. PMID 30052206